CLINICAL TRIAL: NCT05052619
Title: A Prospective, Randomized Clinical Trial to Treat Intra-abdominal Infection Preventively After Pancreatic Surgery Based on Serum Lactate Changes
Brief Title: Preventive Therapy of Postoperative Intra-abdominal Infection Based on Serum Lactate Changes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Lac-infection
Record Dates: First submitted 2021-09-12; First posted 2021-09-22 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Postoperative Infection; Lactate; Antibiotics
Keywords: Serum lactate; Postoperative intra-abdominal infection; Preventive usage; Advanced antibioties; Strategy
MeSH Terms: interventions — sulperazone; Cefmetazole

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Preventive use of advanced antibiotics group (Experimental): Treat patients in this group with advanced preventive usage of antibiocs: Sulperazon 3g q8h, in postoperative days 1-5.
  Interventions: Drug: Preventive use of advanced antibiotics
- Routine group (Other): Treat patients in this group with routine preventive usage of antibiocs: Cefmetazole 1g q12h, in postoperative days 1-3.
  Interventions: Other: Routine

INTERVENTIONS:
Drug: Preventive use of advanced antibiotics — Treat patients in this group with advanced preventive usage of antibiocs: Sulperazon 3g q8h, in postoperative days 1-5.
  Other Names: Sulperazon
  Arms: Preventive use of advanced antibiotics group
Other: Routine — Treat patients in this group with routine preventive usage of antibiocs: Cefmetazole 1g q12h, in postoperative days 1-3.
  Other Names: Cefmetazole
  Arms: Routine group

SUMMARY:
Intra-abdominal infection is one of the most serious complications after pancreatic resection. The preventive use of antibiotics intraoperatively could reduce the incidence rate of postoperative intra-abdominal infection. According to the previous retrospective study, changes of serum lactate level on postoperative day1 could predict the incidence rate of postoperative intra-abdominal infection. This prospective RCT is to further validate and promote the findings and conclusion.

DETAILED DESCRIPTION:
Postoperative intra-abdominal infection is one of the most serious complications after pancreatic resection. Once diagnosed as postoperative intra-abdominal infection, the patient would not only suffer a lot, but also spend much more money and time in hospital. Moreover, subsequent sepsis and septic shock would imperil the patient's life. The preventive use of antibiotics intraoperatively is the key to prevent this complication, but the time, dosage, and choice of the antibiotics are worth discussing. According to the previous work, the investigators found the changes in serum lactate level on postoperative day (POD) 1 could predict postoperative intra-abdominal infection one week before it really happened. The cutoff level of lactate is 3.25mmol/L. Thus, the investigators recommend preventive use of advanced antibiotics for patients who have a peak serum lactate level of >3.250 mmol/L in 24h after pancreatic resection (doi: 10.1007/s00268-021-05987-8. PMID: 33604712).

The investigators would verify the finding in this randomized controlled trial. Patients with peak lactate level >3.250 mmol/L in POD1 and met other inclusion criteria would be recruited and separated into "preventive use of advanced antibiotics group" (experimental group) and "routine group" (control group) randomly. Patients in experimental group would be treated with advanced antibiotics to avoid postoperative intra-abdominal infection. Patients in control group would be treated with routine method (antibiotics with lower levels). To compare the incidence rate of infection and other complications, as well as the payment and other index, the investigators would see if the patients in experimental group could have better prognosis after pancreatic surgery.

ELIGIBILITY:
Inclusion Criteria:

1. treatment by pancreatic resection, including pancreaticoduodenectomy, pancreatosplenectomy, total pancreatectomy, and other variant operations;
2. revival in the intensive care unit (ICU) with standard serum lactate elution treatments after surgery instead of the operation room or general ward;
3. availability of complete preoperative, intraoperative, and postoperative data;
4. the peak serum lactate level in 24 hours after surgery >3.250 mmol/L.

Exclusion Criteria:

1. a history of surgical treatment of any upper abdominal lesions before the current hospital admission;
2. the minimum mean arterial pressure <65 mmHg during the operation;
3. without written informed consents for the perioperative situation and related studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 297 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of postoperative intra-abdominal infection | in 30 days after surgery
  The incidence rate of postoperative intra-abdominal infection is expected to be lower in experimental group than control group

SECONDARY OUTCOMES:
The amount of white blood cell | postoperative days 1, 3, 5, 7, 14, 21, 28
  It is expected to be lower in experimental group than in control group
The level of procalcitonin | postoperative days 1, 3, 5, 7, 14, 21, 28
  It is expected to be lower in experimental group than in control group
The level of C-reactive protein | postoperative days 1, 3, 5, 7, 14, 21, 28
  It is expected to be lower in experimental group than in control group
The level of interleukin | postoperative days 1, 3, 5, 7, 14, 21, 28
  It is expected to be lower in experimental group than in control group
The level of tumor necrosis factor α | postoperative days 1, 3, 5, 7, 14, 21, 28
  It is expected to be lower in experimental group than in control group

CONTACTS AND LOCATIONS:
Overall Officials: Yatong Li, MD, Study Director — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Li Y, Chen L, Xing C, Ding C, Zhang H, Wang S, Long Y, Guo J, Liao Q, Zhang T, Zhao Y, Dai M. Changes in Serum Lactate Level Predict Postoperative Intra-Abdominal Infection After Pancreatic Resection. World J Surg. 2021 Jun;45(6):1877-1886. doi: 10.1007/s00268-021-05987-8. Epub 2021 Feb 18. PMID 33604712
- See also: Previous work of this RCT: the retrospective study — http://pubmed.ncbi.nlm.nih.gov/33604712/